CLINICAL TRIAL: NCT02884817
Title: The Plaque- and Gingivitis Inhibiting Capacity of a Commercially Available Mouthwash Containing Essential Oils and Ethyl Lauroyl Arginate: A Parallel, Split-mouth, Double Blind, Randomized, Placebo-controlled Clinical Study
Brief Title: Essential Oil+ELA, Plaque and Gingivitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oslo (Other)
Responsible Party: Principal Investigator, Hans Ragnar Preus, Professor, University of Oslo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: REK2015/417
Record Dates: First submitted 2016-08-22; First posted 2016-08-31 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-08

CONDITIONS: Dental Plaque; Gingivitis
MeSH Terms: conditions — Dental Plaque; Gingivitis | interventions — Water

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Listerine prof.gum.ther (Experimental): The test solution was the commercially available mouthwash product EOELA that contains essential oils and ELA in 21.6% alcohol (Listerine Professional Gum Therapy®, Johnson & Johnson,USA).
  Intervention; Rinsing 30 sec with test solution twice daily for 21 days
  Interventions: Drug: Experimental: essential oils and ELA
- 21.6% hydroalcoholic (Placebo Comparator): a hydro-alcohol solution made from 96% ethanol diluted with sterilized water to the final concentration of 21.6%.
  Intervention: Rinsing 30 sec with placebo comparator twice daily for 21 days
  Interventions: Other: Placebo
- Plain sterile water (Sham Comparator): Plain sterile water.
  Intervention: Rinsing 30 sec with sham comparator twice daily for 21 days
  Interventions: Other: Water

INTERVENTIONS:
Drug: Experimental: essential oils and ELA — The participants were instructed to insert the tooth guard in Q1 every time they brushed their teeth and to perform a mechanical oral hygiene routine twice a day in the three other quadrants. After brushing properly, they were instructed to rinse for 30s with water before removing the tooth guard. And then rinse again for 30s with water without the mouth guard. Following this procedure the participants rinsed, as instructed, with the Experimental solution, Listerine Gum Therapy. This oral hygiene routine was repeated for 21d.
  Other Names: Listerine Professional Gum Therapy®, Johnson & Johnson,USA
  Arms: Listerine prof.gum.ther
Other: Placebo — The participants were instructed to insert the tooth guard in Q1 every time they brushed their teeth and to perform a mechanical oral hygiene routine twice a day in the three other quadrants. After brushing properly, they were instructed to rinse for 30s with water before removing the tooth guard. And then rinse again for 30s with water without the mouth guard. Following this procedure the participants rinsed, as instructed, with the 21.6% hydroalcoholic solution. This oral hygiene routine was repeated for 21d.
  Other Names: 21.6% hydroalcoholic
  Arms: 21.6% hydroalcoholic
Other: Water — The participants were instructed to insert the tooth guard in Q1 every time they brushed their teeth and to perform a mechanical oral hygiene routine twice a day in the three other quadrants. After brushing properly, they were instructed to rinse for 30s with water before removing the tooth guard. And then rinse again for 30s with water without the mouth guard. Following this procedure the participants rinsed, as instructed, with the sterile water, sham comparator. This oral hygiene routine was repeated for 21d.
  Other Names: Sham Comparator
  Arms: Plain sterile water

SUMMARY:
A commercially available mouth rinse with ethyl lauroyl arginate and essential oils claims to have enhanced antimicrobial properties as compared to the traditional essential oil products. The aim of the present study was to compare the plaque and gingivitis inhibiting effect of the commercial product containing essential oils with ethyl lauroyl arginate with one placebo and one negative control in a modified experimental gingivitis model. In three groups of healthy volunteers, experimental gingivitis was induced and monitored over 21 days, simultaneously treated with the commercial test solution, 21.6% hydro-alcohol solution and sterile water respectively. The maxillary right quadrant of each individual received mouthwash only, whereas the maxillary left quadrant was subject to both rinsing and mechanical oral hygiene. Compliance and side effects were monitored at day 7, 14, and 21. Plaque and gingivitis scores were obtained at baseline and at day 21.

DETAILED DESCRIPTION:
Mouthrinses containing essential oils in 21% - 26% alcohol are claimed to be potent inhibitors of plaque formation, although a recently published study suggests otherwise.

Recently, a new product in this series of mouthwashes was introduced in which an additional antimicrobial agent, Ethyl Lauroyl Arginate, derived from lauric acid and arginine had been added to the standard essential oils and alcohol. Ethyl Lauroyl Arginate acts as a cationic surfactant and has a wide spectrum of activities against Gram positive and - negative bacteria, yeasts and fungi and acts by modifying the permeability of membranes. Ethyl Lauroyl Arginate is used as a multi-functional component in formulations of cosmetic and toiletry products, claiming to act as an anti-static agent and a surfactant with antimicrobial properties. The Scientific Committee on Consumer Safety, has evaluated the safety and use of the ingredient and considered Ethyl Lauroyl Arginate as a safe product when used up to a maximum concentration of 0,15 % in oral dental products. The manufacturer of Essential Oils with Ethyl Lauroyl Arginate claims that Ethyl Lauroyl Arginate prevents the formation of biofilms, and represents a totally new way to combat biofilm-diseases like caries, gingivitis and periodontitis. Moreover, the manufacturer announces that the product reduces plaque colonization of dental surfaces with up to 42.6% and bleeding with up to 50.9% in 4 weeks.

Few or no clinical studies of this new mouthwash have been published, although some informational material is cited in marketing pamphlets.

Thus, the Aim of the present study was to test the clinical plaque- and gingivitis inhibiting capacity of Essential Oils with Ethyl Lauroyl Arginate, with or without mechanical oral hygiene, using a modified experimental gingivitis model, with 21.6 % hydroalcoholic and sterile water as controls.

The HYPOTHESIS was that the test solution was equally effective in preventing dental plaque as the placebo solution in the Experimental gingivitis model.

The present study was designed as a parallel, split-mouth, double masked, randomized, placebo-controlled clinical study. The experimental gingivitis model, with the modifications by Preus et al. was used to induce gingival inflammation under supervised conditions throughout the study. The study was approved by the Regional Committee for Medical Research Ethics, South East Norway, in 2015 and follows the Consort 2010 guidelines.

The study population comprised seventy-four dental, medical, and dental hygienist students, as well as a few clinical teachers, who volunteered to participate in the project. An information meeting was arranged for the volunteers prior to the start of the study, through which the participants received information about oral rinsing products in general and Ethyl Lauroyl Arginate/Essential Oils with Ethyl Lauroyl Arginate products as well as information on the study ahead, in particular. Fifteen subjects withdrew for personal reasons at this time, mostly because they became aware that they could not brush their teeth in the 1st quadrant for 21 days, resulting in fifty-nine participants signing the informed consent form. Mean age was 25 +/- 3.2yr and 78% were females. The study period was 21days, not comprising any special academic, religious or ethnic feasts or events that could jeopardize the collective behavior of the study population. All information, administration and data collection was performed at the Department of Periodontology, Institute of Clinical Odontology, Faculty of Dentistry, University of Oslo, Norway.

Inclusion criteria & Exclusion criteria are listed under "inclusion and Exclusion criteria" below.

The test solution was the commercially available mouthwash product Essential Oils with Ethyl Lauroyl Arginate that contains essential oils and Ethyl Lauroyl Arginate in 21.6% alcohol . The first control was the true placebo solution; a hydro-alcohol solution made from 96% ethanol diluted with sterilized water to the final concentration of 21.6%. The second control solution, plain sterilized water, was used as the negative control because this has been used as control in most studies testing the effect of Ethyl Lauroyl Arginate products. Both control solutions were enriched with 0.2% Fluorid in order to prevent development of early carious lesions during the course of the study. The test solution was not fluoridated since it could change the activity of the active ingredients. The three solutions were filled in identical, labeled (1,2 or 3) bottles.

Randomization was carried out using a computer generated random allocation table assigning the participants to the three study groups with 20 test subjects in each of groups 2 and 3. Group 1 contained 19 participants. They were all carefully instructed to rinse for 30 seconds twice a day with the content of their designated mouthwash. 30 seconds was recommended by the manufacturer for the test solution and was therefore recommended for the controls as well. The statistician performed the randomization whereas the project leader distributed the rinsing solutions and instructions after a list generated as described.

Setting the baseline dental plaque score to zero was done by giving all participants a professional tooth cleaning with rubber cup, pumice paste and dental floss prior to the start of the study on the first day of the study period. Passing baseline, the participants were given their test solution and subsequently instructed to rinse, supervised by the project leader (there and then), as described above with the allocated test solution. This was done since Ethyl Lauroyl Arginate is claimed to be an inhibitor of biofilm formation, and should therefore be applied immediately following the removal of the biofilm. Individual plastic tooth guards had been produced to fit the teeth in the upper right quadrant of each participant prior to baseline. Together with this individual tooth guard, the participants were given identical prophylaxis packs containing a medium texture tooth brush, inter-dental floss and dentifrice. They were instructed to substitute their daily oral hygiene remedies with the ones given to them, and attach the tooth guard to the toothbrush, with a provided rubber string, initially and after use so that the tooth guard always was remembered when using the brush.

The participants were instructed to insert the tooth guard in Quadrant 1 every time they brushed their teeth and to perform a mechanical oral hygiene routine twice a day in the three other quadrants. After brushing properly, they were instructed to rinse for 30 seconds with water before removing the tooth guard. And then rinse again for 30 seconds with water without the mouth guard. Following this procedure the participants rinsed, as instructed, with the solution they randomly had been assigned. This oral hygiene routine was repeated for 21 days. The study design and stringency of logistics ensured that the study participants served as their own controls, as one quadrant was exposed to chemical rinsing only (quadrant 1) and the upper left quadrant (Quadrant 2) received traditional tooth brushing and inter-dental cleaning in addition to the chemical rinsing. Following the last scoring at day 21, the participants received professional tooth cleaning after scoring and before ending the study.

A team of four people were trained in the procedure of informing participants, receiving the test persons for evaluation, questionnaire and clinically monitoring them at all visits. The principal investigator and project managers managed all contact with the participants outside the scoring room. In between appointments the project team kept in touch with the test persons by text messaging and e-mail. The success of this service was evident by zero no-shows at the clinic, as was the case also in the previous studies with this design.

Preceding every examination, the project managers interviewed each participant about compliance and received verbal complaints and descriptions of subjective side-effects. Before entering the scoring room ordered the participants to refrain from any conversation with the scoring scientists inside. The recorders had been instructed likewise.

In the scoring room, two researchers obtained the clinical data. At days 7 and 14 the clinical recordings was based on clinical appearance of adverse effects of the respective solutions. Moreover, these visits were also thought to be important in following the protocol for all participants. At day 21 the plaque index (primary endpoint) and secondary endpoint gingival index (secondary endpoint) were recorded on the mesial, buccal, distal and palatal aspects of teeth 16, 15, 14, 13 and 23, 24, 25, 26. Adverse events like discoloration observed during the clinical examination (yes/no) and clinically visible oral mucosal reactions were registered. In addition, Quigley and Hine plaque index; the Turesky modification, was registered following the above scoring method and dying the Quadrant 1 and Quadrant 2. All clinical registrations were performed by the same experienced periodontist, leaving her colleague to register recordings on especially designed charts. The clinical crew was kept blind to the group allocation of the participants at all times, as the only one that had access to the code-book was the statistician who did not participate in the clinical events.

Statistical analyses The total number of participants was 59, with 19 subjects in group 1, and 20 subjects in group 2 and 3 (using a two-sided t-test with 5% significance level); the test power to detect a true mean difference in Gingival - and Plaque index was above 80%. This power analysis was based on the variable delta plaque, meaning the difference in mean plaque between 1st and 2nd quadrant (test minus control quadrant). When comparing mean variable delta plaque in two groups, a two-sided independent samples t-test was used, with 5% significance level. In the present study sample size was 15 patients in each group. Average standard deviation of DP in the three groups was 0.40. It may be shown that the test power to detect a mean difference of at least 0.40 in the present study when comparing two groups was 78%. As 80% test power is generally considered acceptable in clinical studies and the difference in mean variable Delta Plaque between group 3 and group 1 was 0.49, the above calculation suggests that our study has acceptable test power.

Interval estimates of primary efficacy variables were constructed using 95% as the level of confidence and an overall significance level of 5% was used in the statistical tests. All tests were performed two-sided. The statistical analyses were conducted using the software of Statistical Package for the Social Sciences (SPSS) for Windows, Version 16.0. The difference between groups at day 7, 14 and 21 were tested using an independent samples t-test.

One-way Anova analysis was not used when analyzing the outcome variables, because we considered it most interesting to compare the Alcohol - (group 2) and the Essential Oils with Ethyl Lauroyl Arginate - (group 3) with the reference water group (group 1). The distributions of the outcome variables were checked in hindsight, and found to be sufficiently close to the normal distribution to allow for the use of a t-test.

ELIGIBILITY:
Inclusion Criteria:

healthy subjects from both gender snon-smoking aged 20-55yr having at least three of the following teeth in maxillary right and left quadrant: the canine, 1st bicuspid, 2nd bicuspid, 1st molar, healthy gingiva and periodontium.

Exclusion Criteria:

pregnancy lactation any chronic diseases clinical signs or symptoms of acute infection in the oral cavity any prescribed or non-prescription systemic or topical medication except oral contraceptives clinical parameters judged as unacceptable by the principle investigator use of systemic antibiotics the last 3 months prior to the start of the study history of alcohol or drug abuse participation in other clinical studies in the last 4weeks

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2015-09; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Plaque index (Silness & Loe 1964) | 21 days
  0= No plaque
  1. A film of plaque adhering to the free gingival margin and adjacent area of the tooth. The plaque may be seen in situ only after application of disclosing solution or by using the probe on the tooth surface.
  2. Moderate accumulation of soft deposit s within the gingival pocket, or the tooth and gingival margin which can be seen with the naked eye.
  3. Abundance of soft matter within the gingival pocket and/or on the tooth and gingival margin.

SECONDARY OUTCOMES:
The gingival index (GI) (Løe & Silness 1963) | 21 days
  0 No inflammation.
  1. Mild inflammation, slight change in color, slight edema, no bleeding on probing.
  2. Moderate inflammation, moderate glazing, redness, bleeding on probing.
  3. Severe inflammation, marked redness and hypertrophy, ulceration, tendency to spontaneous bleeding.

OTHER OUTCOMES:
Ill or side effects | 21 days
  All reported side subjective side effects like "loss of taste", "numbness ...
Objective observation of Discoloration of teeth | 21 days
  Clinical observation of discoloration; Slight to obvious

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Periodontology, Institute of Clinical Odontology, Dental Faculty, University of Oslo, Oslo, Oslo County, Norway

IPD SHARING:
Plan to Share IPD: Yes
Via scientific journals

REFERENCES:
- [Background] McCullough MJ, Farah CS. The role of alcohol in oral carcinogenesis with particular reference to alcohol-containing mouthwashes. Aust Dent J. 2008 Dec;53(4):302-5. doi: 10.1111/j.1834-7819.2008.00070.x. PMID 19133944
- [Background] Van Leeuwen MP, Slot DE, Van der Weijden GA. Essential oils compared to chlorhexidine with respect to plaque and parameters of gingival inflammation: a systematic review. J Periodontol. 2011 Feb;82(2):174-94. doi: 10.1902/jop.2010.100266. Epub 2010 Nov 2. PMID 21043801
- [Background] Preus HR, Koldsland OC, Aass AM, Sandvik L, Hansen BF. The plaque- and gingivitis-inhibiting capacity of a commercially available essential oil product. A parallel, split-mouth, single blind, randomized, placebo-controlled clinical study. Acta Odontol Scand. 2013 Nov;71(6):1613-9. doi: 10.3109/00016357.2013.782506. Epub 2013 May 3. PMID 23638764
- [Background] Hawkins DR, Rocabayera X, Ruckman S, Segret R, Shaw D. Metabolism and pharmacokinetics of ethyl N(alpha)-lauroyl-L-arginate hydrochloride in human volunteers. Food Chem Toxicol. 2009 Nov;47(11):2711-5. doi: 10.1016/j.fct.2009.07.028. Epub 2009 Aug 3. PMID 19651183
- [Background] Gallob JT, Lynch M, Charles C, Ricci-Nittel D, Mordas C, Gambogi R, Revankar R, Mutti B, Labella R. A randomized trial of ethyl lauroyl arginate-containing mouthrinse in the control of gingivitis. J Clin Periodontol. 2015 Aug;42(8):740-747. doi: 10.1111/jcpe.12428. Epub 2015 Aug 15. PMID 26087864
- [Background] LOE H, THEILADE E, JENSEN SB. EXPERIMENTAL GINGIVITIS IN MAN. J Periodontol (1930). 1965 May-Jun;36:177-87. doi: 10.1902/jop.1965.36.3.177. No abstract available. PMID 14296927
- [Background] Preus HR, Aass AM, Hansen BF, Moe B, Gjermo P. A randomized, single-blind, parallel-group clinical study to evaluate the effect of soluble beta-1,3/1,6-glucan on experimental gingivitis in man. J Clin Periodontol. 2008 Mar;35(3):236-41. doi: 10.1111/j.1600-051X.2007.01183.x. PMID 18269662
- [Background] Altman DG. Clinical Trials. Practical statistics for medical research. London:Chapman & Hall/CRC, 1991;456.
- [Background] QUEIROZ DR, MORDAS CJ, MARTINEZ MD, SHANG H, GAMBOGI RJ. Examination of Ethyl-Lauroyl-Arginate-HCl (LAE) Deposition on a Model Enamel Surface. IADR Abstract and Programme 2015; Abstr 0559, Boston March 12th, 2015
- [Background] http://www.google.com/patents/US20040258632 *
- [Background] https://www.foodstandards.gov.au/code/applications/documents/AR_A1015.pdf *
- [Background] http://ec.europa.eu/health/ph_risk/committees/04_sccp/docs/sccp_o_017.pdf *
- [Background] http://www.lamirsa.com/mirenat/pdf/03-PCT.pdf
- [Background] http://ec.europa.eu/health/scientific_committees/consumer_safety/docs/sccs_o_138.pdf
- [Background] http://www.nature.com/bdj/journal/v218/n6/full/sj.bdj.2015.234.html
- [Background] http://barkerpr.com/2014/05/advanced-defence-gum-treatment/
- [Background] SILNESS J, LOE H. PERIODONTAL DISEASE IN PREGNANCY. II. CORRELATION BETWEEN ORAL HYGIENE AND PERIODONTAL CONDTION. Acta Odontol Scand. 1964 Feb;22:121-35. doi: 10.3109/00016356408993968. No abstract available. PMID 14158464
- [Background] LOE H, SILNESS J. PERIODONTAL DISEASE IN PREGNANCY. I. PREVALENCE AND SEVERITY. Acta Odontol Scand. 1963 Dec;21:533-51. doi: 10.3109/00016356309011240. No abstract available. PMID 14121956
- [Background] QUIGLEY GA, HEIN JW. Comparative cleansing efficiency of manual and power brushing. J Am Dent Assoc. 1962 Jul;65:26-9. doi: 10.14219/jada.archive.1962.0184. No abstract available. PMID 14489483
- [Background] Turesky S, Gilmore ND, Glickman I. Reduced plaque formation by the chloromethyl analogue of victamine C. J Periodontol. 1970 Jan;41(1):41-3. doi: 10.1902/jop.1970.41.41.41. No abstract available. PMID 5264376
- [Background] Vatne JF, Gjermo P, Sandvik L, Preus HR. Patients' perception of own efforts versus clinically observed outcomes of non-surgical periodontal therapy in a Norwegian population: an observational study. BMC Oral Health. 2015 May 17;15:61. doi: 10.1186/s12903-015-0037-3. PMID 25981528
- [Background] Preus HR, Dahlen G, Gjermo P, Baelum V. Microbiologic Observations After Four Treatment Strategies Among Patients With Periodontitis Maintaining a High Standard of Oral Hygiene: Secondary Analysis of a Randomized Controlled Clinical Trial. J Periodontol. 2015 Jul;86(7):856-65. doi: 10.1902/jop.2015.140620. Epub 2015 Mar 12. PMID 25762359
- [Background] Guha N, Boffetta P, Wunsch Filho V, Eluf Neto J, Shangina O, Zaridze D, Curado MP, Koifman S, Matos E, Menezes A, Szeszenia-Dabrowska N, Fernandez L, Mates D, Daudt AW, Lissowska J, Dikshit R, Brennan P. Oral health and risk of squamous cell carcinoma of the head and neck and esophagus: results of two multicentric case-control studies. Am J Epidemiol. 2007 Nov 15;166(10):1159-73. doi: 10.1093/aje/kwm193. Epub 2007 Aug 30. PMID 17761691
- [Background] Werner CW, Seymour RA. Are alcohol containing mouthwashes safe? Br Dent J. 2009 Nov 28;207(10):E19; discussion 488-9. doi: 10.1038/sj.bdj.2009.1014. PMID 19942865
- [Derived] Valor LO, Norton IKR, Koldsland OC, Aass AM, Grjibovski AM, Preus HR. The plaque and gingivitis inhibiting capacity of a commercially available mouthwash containing essential oils and ethyl lauroyl arginate. A randomized clinical trial. Acta Odontol Scand. 2018 May;76(4):241-246. doi: 10.1080/00016357.2017.1412499. Epub 2017 Dec 7. PMID 29216779